CLINICAL TRIAL: NCT05985616
Title: Effects of High Intensity Resistance Training on Physical Function in Possible Sarcopenia Cases
Brief Title: High Intensity Resistance Training and Possible Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC01549 Shanza Nisar
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): High intensity (80-85% of 1RM) will be administered at alternative days for 16 weeks.
  The exercise will have three phases; Phase I consists of 2-3 sets of 8-15 repetitions, Phase II will follow the single set approach and Phase III will have the Superset approach.
  The following activities will be incorporated via resistance training: latissimus front pulleys, rowing, back extension, inverse fly, bench press, shoulder press, lateral raises, butterfly with extended arms, crunches, leg presses, leg extension and curls, leg adduction, abduction.
  Interventions: Other: High Intensity Resistance Training
- Group B (No Intervention): No intervention will be provided in this group. The participants in this group will follow their usual daily activities.

INTERVENTIONS:
Other: High Intensity Resistance Training — High intensity resistance training will be performed 3 times a day for sixteen weeks
  Arms: Group A

SUMMARY:
Studies conducted so far added the dietary supplements along with resistance training as an intervention, we could not determine whether the observed effects of the intervention were due to the training program and/or dietary supplements.

DETAILED DESCRIPTION:
This study will investigate the effects of high intensity resistance training solely in the possible sarcopenia cases which has not done before, to author's knowledge. Furthermore this study will help clinicians to individualize and optimize the therapy for specific patient subgroups, improve the potential of this therapy to improve human function and well being, facilitate timely interventions in community healthcare and prevention settings, which will contribute to higher awareness of sarcopenia prevention and interventions in diverse health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age more than 60 years
* Possible sarcopenia cases as defined by Asian Working Group for Sarcopenia (Handgrip strength: Male less than 26kg and Female less than 18kg, 5 time chair stand test more than/equals to 12 seconds)

Exclusion Criteria:

* Orthopedic surgery in last one year
* Neurological disorders like stroke etc
* History of recent fractures
* Metabolic disorders like DM etc
* Actively involved in exercise programs
* Cognitive impairment that could confound the assessment
* Wheelchair or bed bound individuals

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Hand Dynamometer | 16 weeks
  it used to measure the hand grip strength. the test-retest reliability is 0.91 and 0.95 with excellent reliability. The assessment will be made at baseline, week 8 and 16
Short performance physical battery | 16 Week
  an objective assessment tool for evaluating lower extremity functioning in older persons. the test-retest reliability is 0.87. It was used to measure at baseline, week 8 and 16

SECONDARY OUTCOMES:
FRAIL | 16 week
  The questionnaire aims at fatigue, resistance, ambulation, illness and loss of weight. It is a self reported questionnaire. The sensitivity of FRAIL is 85.8% and a specificity of 80.6%.
  The test will be measured at baseline, week 8 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Abbas Institute of Medical Sciences, Muzaffarabad, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kemmler W, Kohl M, Frohlich M, Jakob F, Engelke K, von Stengel S, Schoene D. Effects of High-Intensity Resistance Training on Osteopenia and Sarcopenia Parameters in Older Men with Osteosarcopenia-One-Year Results of the Randomized Controlled Franconian Osteopenia and Sarcopenia Trial (FrOST). J Bone Miner Res. 2020 Sep;35(9):1634-1644. doi: 10.1002/jbmr.4027. Epub 2020 Apr 28. PMID 32270891
- [Background] Singh M, Stewart R, White H. Importance of frailty in patients with cardiovascular disease. Eur Heart J. 2014 Jul;35(26):1726-31. doi: 10.1093/eurheartj/ehu197. Epub 2014 May 26. PMID 24864078
- [Background] Abdul-Hameed U, Rangra P, Shareef MY, Hussain ME. Reliability of 1-repetition maximum estimation for upper and lower body muscular strength measurement in untrained middle aged type 2 diabetic patients. Asian J Sports Med. 2012 Dec;3(4):267-73. doi: 10.5812/asjsm.34549. PMID 23342225